CLINICAL TRIAL: NCT02619656
Title: Insufflation With Carbon Dioxide Reduces Pneumoperitoneum After Percutaneous Endoscopic Gastrostomy (PEG): A Randomized Controlled Trial
Brief Title: A Trial of Supplemental CO2 Versus Room Air in Percutaneous Endoscopic Gastrostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, John C. Fang, M.D., Chief, Division of Gastroenterology, Hepatology and Nutrition, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 55102
Record Dates: First submitted 2015-11-10; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Pneumoperitoneum
Keywords: PEG; CO2 insufflation; Room Air insufflation; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Patients randomized to insufflation with CO2.
  Intervention: CO2 Insufflation with CO2Efficient Endoscopic Insufflator on managed flow setting at 3.4 L/min
  Interventions: Procedure: CO2 insufflation
- Control (Active Comparator): Patients randomized to insufflation with ambient air.
  Intervention: Ambient air insufflation with Evis Exera 111 CLV-190 on medium air flow setting 0.68 L/min
  Interventions: Procedure: Ambient air insufflation

INTERVENTIONS:
Procedure: CO2 insufflation — Patients were randomized to insufflation with CO2.
  Other Names: CO2Efficient Endoscopic Insufflator on flow setting 3.4L/min
  Arms: Treatment
Procedure: Ambient air insufflation — Patients were randomized to insufflation with ambient air.
  Other Names: Evis Exera 111 CLV-190 on medium air flow setting 0.68L/min
  Arms: Control

SUMMARY:
The investigators hypothesize that using carbon dioxide for PEG placement versus using room air will decrease post-procedure pneumoperitoneum as well as improve post-procedure bloating/pain, and waist circumference.

DETAILED DESCRIPTION:
Background and study aims: Pneumoperitoneum following PEG placement has been reported in up to 60% of cases, and while usually benign and self-limited, it can lead to evaluation for suspected perforation. This study was designed to determine whether using CO2 compared to ambient air for insufflation during PEG reduces post-procedure pneumoperitoneum.

Patients and Methods: Prospective, double blind, randomized trial of 35 consecutive patients undergoing PEG at a single academic medical center. Patients were randomized to insufflation with CO2 or ambient air. Primary outcome was pneumoperitoneum determined by left-lateral decubitus abdominal x-rays 30 min after PEG placement. Secondary endpoints included abdominal distention, pain, and bloating.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 and need a percutaneous endoscopic gastrostomy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Post-procedure pneumoperitoneum | left-lateral decubitus abdominal x-rays 30 min after PEG placement.
  Frequency of post pneumoperitoneum determined by left-lateral decubitus abdominal x-rays 30 min after PEG placement.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Murphy, MD, Study Chair — University of Utah SOM; John C Fang, MD, Principal Investigator — University of Utah SOM
Locations (1):
- University of Utah SOM, Salt Lake City, Utah, United States